CLINICAL TRIAL: NCT01845376
Title: Postoperative Clinical Outcomes and Inflammatory Markers After Inguinal Hernia Repair With Local or Spinal or General Anesthesia: A Randomized Trial
Brief Title: Local or Regional or General Anesthesia for Hernia Repair: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mingkwan Wongyingsinn, MD (Other)
Responsible Party: Sponsor-Investigator, Mingkwan Wongyingsinn, MD, Assistant professor, Doctor, Siriraj Hospital
Organization: Siriraj Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIRB035
Record Dates: First submitted 2013-04-26; First posted 2013-05-03 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Hernia; Anesthetics Adverse Reaction; Inflammation
Keywords: Inflammatory Markers after Inguinal Hernia Repair; Anesthetic technique for hernia repair
MeSH Terms: conditions — Hernia; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- local anesthesia group (Experimental): In the local anesthesia group, patients will receive local anesthesia similar to that described by Amid et al. except that 1% lidocaine with adrenaline (1:200,000) will be used instead of a mixture of lidocaine and bupivacaine. Surgeons will be taught to do the local anesthetic technique in a standardized manner.
  Interventions: Procedure: local anesthesia group
- spinal anesthesia group (Experimental): In the spinal anesthesia group, patients will be positioned in the lateral position and a Whitacre 25 G needle will be inserted at L3-4 intervertebral space and then heavy bupivacaine 0.5% 15 mg will be injected. Sensory block (T4 and below dermatomes) to cold and pinprick will be tested before starting operation. An incremental dose containing 1 mg of midazolam and 25 mcg of fentanyl will be intravenously given if patients in the LA and SA group require.
  Interventions: Procedure: spinal anesthesia group
- general anesthesia group (Experimental): In the general anesthesia group, patients will be induced with propofol 2 mg/kg and fentanyl 1.5 µg /kg. They are then allowed to breathe spontaneously with sevoflurane 2% to 2.5% in a mixture of 60% oxygen through a laryngeal mask. End-tidal concentration of sevoflurane will be adjusted to keep end-tidal sevoflurane 1MAC. Supplemental doses of 25 µg of fentanyl will be administered if intraoperative heart rate and blood pressure are greater than 20% of baseline.
  Interventions: Procedure: general anesthesia group

INTERVENTIONS:
Procedure: local anesthesia group — Patients will receive local anesthesia similar to that described by Amid et al. except that 1% lidocaine with adrenaline (1:200,000) will be used instead of a mixture of lidocaine and bupivacaine.
  Other Names: LA group
  Arms: local anesthesia group
Procedure: spinal anesthesia group — Patients will be positioned in the lateral position and a Whitacre 25 G needle will be inserted at L3-4 intervertebral space and then heavy bupivacaine 0.5% 15 mg will be injected.
  Other Names: SA group
  Arms: spinal anesthesia group
Procedure: general anesthesia group — Patients will be induced with propofol 2 mg/kg and fentanyl 1.5 µg /kg. They are then allowed to breathe spontaneously with sevoflurane 2% to 2.5% in a mixture of 60% oxygen through a laryngeal mask. End-tidal concentration of sevoflurane will be adjusted to keep end-tidal sevoflurane 1MAC. Supplemental doses of 25 µg of fentanyl will be administered if intraoperative heart rate and blood pressure are greater than 20% of baseline.
  Other Names: GA group
  Arms: general anesthesia group

SUMMARY:
This present randomized trial is designed to evaluate the postoperative pain,inflammatory marker, postoperative analgesic medication, length of hospital stay and the modifications of inflammatory mediators in patients undergoing inguinal hernia repair using local, spinal or general anesthesia.

DETAILED DESCRIPTION:
After approval by Siriraj Institutional Review Board, a prospective randomized study in patients scheduled to undergo elective unilateral inguinal hernia repair at Siriraj Hospital will be undertaken. Patients, ASA I-III, greater than 18 years old will be approached in the outpatient surgical department and recruited in this study. Informed written consent will be obtained from each of them. Exclusion criteria are allergy to any medication used this study, femoral hernia, recurrent hernia, bilateral hernia, bleeding abnormalities, severe hepatic, renal or cardiovascular disease, chronic use of opioid, history of using steroidal or nonsteroidal anti-inflammatory drugs in the past 6 months, inability to communicate in Thai or to understand the purpose of the study.

Anesthesia and surgical procedure

All patients will be admitted one day before operation as routine and receive no premedication. Patients will be randomly allocated in the morning of the operation to receive one of the three anesthetic techniques: local anesthesia (LA), spinal anesthesia (SA) or general anesthesia (GA) for their inguinal hernia repair. The randomization process will be done by the use of a computer-generated number sealed in a brown envelope. All the patients will undergo standardized inguinal hernia repairs by three surgeons, A Trakarnsanga; V Chinsawangtanakul; T Akaraviputh, who agree to follow a precise protocol using Lichtenstein technique as described by Amid.

In the LA group, patients will receive local anesthesia similar to that described by Amid et al. except that 1% lidocaine with adrenaline (1:200,000) will be used instead of a mixture of lidocaine and bupivacaine. Surgeons will be taught to do the local anesthetic technique in a standardized manner.

In the SA group, patients will be positioned in the lateral position and a Whitacre 25 G needle will be inserted at L3-4 intervertebral space and then heavy bupivacaine 0.5% 15 mg will be injected. Sensory block (T4 and below dermatomes) to cold and pinprick will be tested before starting operation. An incremental dose containing 1 mg of midazolam and 25 mcg of fentanyl will be intravenously given if patients in the LA and SA group require.

In the GA group, patients will be induced with propofol 2 mg/kg and fentanyl 1.5 µg /kg. They are then allowed to breathe spontaneously with sevoflurane 2% to 2.5% in a mixture of 60% oxygen through a laryngeal mask. End-tidal concentration of sevoflurane will be adjusted to keep end-tidal sevoflurane 1MAC. Supplemental doses of 25 µg of fentanyl will be administered if intraoperative heart rate and blood pressure are greater than 20% of baseline.

For postoperative analgesia, all groups will receive infiltration 10 ml of 0.5% into the surgical wounds. They will also receive oral acetaminophen two tablets every 6 hours and Arcoxia® (etoricoxib) 60-90 mg daily unless contraindicated for the duration of their hospital stay. Intravenous morphine 1-2 mg will be provided every 4 hours as a breakthrough medication.

For hospital discharge, patients will be allowed to discharge home when they fulfill criteria: obtain and self-administer medications; perform self-care activities; eat an appropriate diet or otherwise manage nutritional needs; follow-up with designated providers.

A blood sample 7 mL will be taken at antecubital vein with aseptic technique, proper decontamination procedures and needle 22-gauge on the preoperative day, at 8 and 24 hours after completion of the surgery. Blood samples will be collected in tubes without anticoagulant to perform interleukin-1 beta (IL-1 beta), IL-6 and IL-10 assays. All blood samples will be centrifuged for 15 min at 1000g. Serum will be stored at -80 °C until performing assay for cytokines. The IL-1 beta, IL-6 and IL-10 will be assessed in the serum with LEGEND MAX Human Interleukin ELISA Kit (Biolegend, USA). Briefly, the quantitative sandwich enzyme immunoassay technique uses monoclonal antibodies specific for IL-1 beta or IL-6 or IL-10. Serum concentrations will be calculated by using regression analysis with standard curves and expressed as picograms per milliliter (pg /ml). All samples will be measured in duplicate, with averages used in the statistical analyses. The minimum detectable concentrations IL-1 beta, IL-6 and IL-10 are 0.5 pg /ml, 1.6 pg /ml and 2 pg /ml, respectively.

All the perioperative data will be collected from patients' chart and filled in case record form by one of the authors. The ward nurses round and the postoperative anesthetic nurses round will follow the care pathway as routine. Patients have no restrictions on activities, and they are encouraged to resume work and normal daily activities as soon as possible. Patients are discharged in accordance with routine at our respective hospital.

The following data will be collected: demographic characteristics, diagnosis, duration of anesthesia and surgery, conversion to other anesthetic techniques or other operations, quality of pain relief, postoperative use of analgesics and amount of analgesic medication, intraoperative and postoperative complications, incidence of postoperative nausea and vomiting (PONV), length of postoperative hospital stay, acute inflammatory markers, patient satisfaction, incidence of complications and readmission rate during 30 days after the operation. Complications are defined as bleeding or hematoma necessitating reoperation or compression bandage, urinary retention that requires catheterization, fever > 38°Celsius requiring medication treatment.

Primary outcomes are postoperative pain at rest and on mobilization at postoperative 8 and 24 as measured with verbal rating score (VRS) from 0 (no pain) to 10 (worst pain). Secondary outcome measures are acute inflammatory markers. Intermediate outcomes include duration of anesthesia and surgery, conversion to other anesthetic techniques, postoperative use of analgesics and amount of analgesic medication, incidence of nausea and vomiting, length of postoperative hospital stay in the unit of hour, patient satisfaction measured with verbal rating score (VRS) from 0 (worst) to 100 (best), incidence of complications and readmission rate during 30 days after the operation.

The primary outcome is postoperative pain on mobilization at 24 after the operation. The sample size is based on two previous studies, which the pain scores of patients having local anesthesia is 5.2 (SD=4.38), spinal anesthesia is 4.0 (SD=2.08) and general anesthesia is 7.2 (SD=1.73), a calculation is done to obtain a type I error of 0.05 and a power of 80% with a balanced Analysis Of Variance test (ANOVA) using nQuery Advisor version 7.0 (Statistical Solutions, Cork, Ireland).2, 4 The calculated sample size per group is 15 patients and the number is increased to 18 patients per groups to include 20% dropouts.

Categorical variables are analyzed by X2 test. Continuous variables are presented as mean and standard deviation (SD) or median and interquartile range (IQR) when data are not normal distribution. Comparison between groups used either ANOVA with Bonferroni's post hoc test or Kruskall Wallis test when data are not normally distributed. All statistical tests are two tailed and P value less than 0.05 is considered significant for all data. Statistical analysis is performed using SPSS version 18 for Windows (SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective unilateral inguinal hernia repair at Siriraj Hospital will be undertaken.
* ASA I-III,
* Age greater than 18 years old

Exclusion Criteria:

* Allergy to any medication used this study,
* Femoral hernia, recurrent hernia, bilateral hernia,
* Bleeding abnormalities,
* Severe hepatic, renal or cardiovascular disease,
* Chronic use of opioid,
* History of using steroidal or nonsteroidal anti-inflammatory drugs in the past 6 months,
* Inability to communicate in Thai or to understand the purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
postoperative pain on mobilization | at postoperative 8 hours
  postoperative pain on mobilization at postoperative 8 hour. postoperative pain is measured with verbal rating score (VRS) from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
acute inflammatory markers (IL-1 beta) | at 8 hours after surgery
  All samples will be measured in duplicate, with averages used in the statistical analyses. The minimum detectable concentrations IL-1 beta, IL-6 and IL-10 are 0.5 pg /ml, 1.6 pg /ml and 2 pg /ml, respectively.
acute inflammatory markers (IL-6) | at 8 hours after surgery
  All samples will be measured in duplicate, with averages used in the statistical analyses.
acute inflammatory markers (IL-10) | at 8 hours after surgery
  All samples will be measured in duplicate, with averages used in the statistical analyses.

OTHER OUTCOMES:
conversion to other anesthetic techniques | at 2 hours after operation
postoperative use of analgesics and amount of analgesic medication | in the period of 24 hours after operation
incidence of complication | 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, MD, MSc, Principal Investigator — Department of Anesthesiology
Locations (1):
- Siriraj hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No